CLINICAL TRIAL: NCT05788510
Title: Pneumococcal Vaccination in Patients with Anti-TNF Alpha Therapy: Status Report on the NOVO Hospital - Pontoise Site
Brief Title: Pneumococcal Vaccination in Patients with Anti-TNF Alpha Therapy
Acronym: TNF-VAX
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD 0423
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-05

CONDITIONS: Pneumococcal Vaccine
Keywords: Pneumococcal vaccine; Immunosupressed patients; Immunization status; Anti-TNF alpha
MeSH Terms: interventions — Pneumococcal Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pneumococcal vaccine: Investigation of vaccination status, for Pneumococcal vaccine , of patients who received anti-TNF alpha therapy
  Interventions: Other: Pneumococcal vaccine

INTERVENTIONS:
Other: Pneumococcal vaccine — Investigation of vaccination status, for Pneumococcal vaccine , of patients who received anti-TNF alpha therapy

SUMMARY:
As the vaccination of immunosuppressed people is insufficiently performed in France, it seems interesting to carry out an evaluation of the situation on the site of the NOVO - Pontoise hospital.

The aim of this study is to assess the status of pneumococcal vaccination in patients at the NOVO hospital - Pontoise site, who have received anti-TNF alpha therapy.

DETAILED DESCRIPTION:
Immunosuppressed patients are at risk of infections, sometimes severe with life-threatening consequences. Some of these are vaccine-preventable, notably pneumococcal infections. Specific vaccination recommendations have been published since 2012 by the French High Council for Public Health. However, vaccine coverage is below the desired immunisation objectives for immunosuppressed patients.

As the vaccination of immunosuppressed people is insufficiently performed in France, it seems interesting to carry out an evaluation of the situation on the site of the NOVO - Pontoise hospital, in order to propose, if necessary, measures, in particular a specialised consultation, with the aim of improving the vaccination coverage of this population at risk The aim of this study is to assess the status of pneumococcal vaccination in patients who have received anti-TNF alpha therapy.

ELIGIBILITY:
Inclusion Criteria :

* Patients treated with anti-TNF alpha between 2020 and 2022 at the NOVO Hospital - Pontoise site

Exclusion Criteria :

* Patients with an indication for pneumococcal vaccination who have received a full vaccination regimen prior to the decision to start anti-TNF alpha

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having received anti-TNF alpha treatment between 2020 and 2022 at the NOVO Hospital - Pontoise site
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the prescription of a pneumococcal vaccination (Conjugated or Unconjugated Pneumococcal Vaccine) by doctors practising at the NOVO Hospital - Pontoise site, in patients receiving anti-TNF alpha treatment | At the end of the study, an average of one month
  Presence or absence of a prescription or completion of a complete pneumococcal vaccination (Conjugated Pneumococcal Vaccine 13-valent or Unconjugated Pneumococcal Vaccine 23-valent) recorded in the patient's medical file.

SECONDARY OUTCOMES:
Assessment of the timing of the vaccines (Conjugated Pneumococcal Vaccine 13-valent or Unconjugated Pneumococcal Vaccine 23-valent) in relation to the date of initiation of anti-TNF alpha therapy | At the end of the study, an average of one month
  Number of patients who received a complete pneumococcal vaccination before initiation of treatment and the number of patients who received it after
Assessment of the number of injections prescribed and/or performed (Conjugated Pneumococcal Vaccine 13-valent or Unconjugated Pneumococcal Vaccine 23-valent) for each patient | At the end of the study, an average of one month
  Number of patients who received an incomplete vaccination scheme (1 dose of Conjugated Pneumococcal Vaccine 13-valent or Unconjugated Pneumococcal Vaccine 23-valent).
Evaluation of the prescription or completion of the vaccination according to the characteristics of the patients and their comorbidities. | At the end of the study, an average of one month
  Analysis of the data to identify any significant differences according to the characteristics of the vaccinated and non-vaccinated patients (comorbidities, pathology for which the treatment was introduced .....).
Evaluation of the prescription or completion of the vaccination according to the medical specialty of the prescriber | At the end of the study, an average of one month
  Analysis of the data to identify any significant differences according to the medical specialty of the prescriber.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Christine Trumtel, Principal Investigator — NOVO Hospital
Locations (1):
- Internal Medicine Department - NOVO Hospital - Pontoise site, Pontoise, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: COVARISQ (estimation de la COuverture VAccinale des adultes à RISQues) : taux de vaccination des immunodéprimés en France en 2017 — https://www.em-consulte.com/article/1383294/covarisq-estimation-de-la-couverture-vaccinale-des
- See also: Haut Conseil de Santé Public - Vaccination des personnes immunodéprimées ou aspléniques - Recommandations - Rapport 2012 — https://www.hcsp.fr/explore.cgi/avisrapportsdomaine?clefr=504